CLINICAL TRIAL: NCT03623880
Title: Enhancing Behavioral Treatment for Women With Pelvic Floor Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, James W Griffith, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00207124
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Floor Disorders; Anxiety; Urinary Urgency; Urinary Incontinence; Nocturia; Urinary Frequency/Urgency; Lower Urinary Tract Symptoms; Urinary Hesitancy; Urinary Straining
MeSH Terms: conditions — Pelvic Floor Disorders; Anxiety Disorders; Urinary Incontinence; Nocturia; Lower Urinary Tract Symptoms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (Experimental): This is a type of CBT for emotional distress.
  Interventions: Behavioral: Unified Protocol
- Supportive Therapy (Active Comparator): This is a commonly-used form of all-purpose psychotherapy, often used as a comparator in CBT clinical trials.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Unified Protocol — The unified protocol is a form of cognitive behavior therapy focused on helping the person reduce emotional distress through cognitive changes and behavioral skills. Exercises included confronting emotional-driven behaviors and mindfulness activities.
  Arms: Unified Protocol
Behavioral: Supportive Therapy — Supportive therapy seeks to improve self-esteem, aid the patient with problem solving, and provide structured support using empathetic listening.
  Arms: Supportive Therapy

SUMMARY:
The purpose of this proposal is to test a novel behavioral treatment - Unified Protocol Cognitive-Behavior Therapy (UP-CBT)1 - to enhance quality of life in women with pelvic floor disorders. Emotional distress is treatable using behavioral procedures, and effective treatment would increase women's emotional health and help to reduce urinary symptoms (e.g., incontinence, frequent urination). Women with pelvic floor disorders are often seen in the urogynecology clinic, which makes this setting ideal for offering additional interventions that may improve their quality of life. Unfortunately, many women with pelvic floor disorders may not receive effective behavioral treatment, such as cognitive behavior therapy, because urogynecologists and other medical professionals may not be aware of providers in their community who offer this treatment. The investigators will enhance treatment options by 1) providing evidence for an all-purpose cognitive-behavioral intervention (i.e., UP-CBT), 2) offering treatment in the urogynecology clinic, maximizing convenience, and 3) improving clinical outcomes for these patients.

Specific Aims:

1. To demonstrate that UP-CBT is an effective form of therapy for women with lower urinary tract symptoms.
2. To use baseline characteristics in moderation analyses to determine which women will be most likely to have a good response to therapy.
3. To use mediation analyses to test a possible causal chain of events - Does treatment lead to lower anxiety, which in turn leads to fewer urinary symptoms?

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* Presence of one or more of the following urinary symptoms in past 12 months and currently seeking treatment: frequency, nocturia, urgency, leakage, hesitancy, straining, or dribbling
* Willing and able to provide informed consent
* Anxious presentation and/or history of anxiety
* English speaking
* Willing to defer usual treatment for urinary problems

Exclusion Criteria:

* Blood in the urine, positive urine culture, signs of infection
* Pregnant, or 6 months or less postpartum
* Psychosis, dementia, or other cognitive impairment that would preclude participation
* Recent (within 6 months) pelvic or endoscopic surgery, urethral stricture, pelvic malignancy, current chemotherapy or other cancer therapy, pelvic device or implant complication
* Recent (within 12 months) Botox injection to the bladder or pelvic structures
* Currently in psychotherapy
* Current alcohol or substance use disorder
* Difficulty communicating in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 38 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Anxiety 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of anxiety symptoms. Min T Score = 40.3; Max T Score = 81.6. Raw scores are summed, then converted to T Scores from a lookup table. Higher T scores represent a worse outcome (i.e., greater number of anxiety symptoms).
Urinary Distress Inventory (UDI-6) | 3 months; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of urinary symptoms and bother. Scores are scale scores: mean value of items answered multiplied by 25; min scale score = 0; max scale score = 100. This scale score can be combined with the scale scores of the Pelvic Organ Prolapse Distress Inventory (POPDI-6) and Colorectal-Anal Distress Inventory (CRAD-8) to form the Pelvic Floor Distress Inventory (PFDI-20) summary score: add three scale scores together (range 0 to 300). Higher score indicates worse outcome (i.e., greater urinary symptoms and bother).

SECONDARY OUTCOMES:
Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6) | 3 months; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of pelvic symptoms and bother. Sores are scale scores: mean value of items answered multiplied by 25; min scale score = 0; max scale score = 100. This scale score can be combined with the scale scores of the UDI-6 and CRAD-8 to form the PFDI-20 summary score: add three scale scores together (range 0 to 300). Higher score indicates worse outcome (i.e., greater pelvic symptoms and bother).
Colorectal-Anal distress Inventory 8 (CRAD-8) | 3 months; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of colorectal-anal symptoms and bother. Sores are scale scores: mean value of items answered multiplied by 25; min scale score = 0; max scale score = 100. This scale score can be combined with the scale scores of the POPDI-6 and UDI-6 to form the PFDI-20 summary score: add three scale scores together (range 0 to 300). Higher score indicates worse outcome (i.e., greater colorectal-anal symptoms and bother).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Depression 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of depression symptoms. Min T Score = 41.0; Max T Score = 79.4. Raw scores are summed, then converted to T Scores from a lookup table. Higher T scores represent a worse outcome (i.e., greater number of depressive symptoms).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Physical Function 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of physical function. Min T Score = 22.9; Max T Score = 56.9. Raw scores are summed, then converted to T Scores from a lookup table. Lower T scores represent a worse outcome (i.e., worse physical functioning).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Fatigue 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of fatigue. Min T Score = 33.7; Max T Score = 75.8. Raw scores are summed, then converted to T Scores from a lookup table. Higher T scores represent a worse outcome (i.e., greater fatigue).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Sleep Disturbance 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of sleep quality and disturbance. Min T Score = 32.0; Max T Score = 73.3. Raw scores are summed, then converted to T Scores from a lookup table. Higher T scores represent a worse outcome (i.e., greater sleep disturbance).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Ability to Participate in Social Roles and Activities 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of social role function. Min T Score = 27.5; Max T Score = 64.2. Raw scores are summed, then converted to T Scores from a lookup table. Lower T scores represent a worse outcome (i.e., greater difficulty participating in social roles/activities).
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 - Profile V2.0: Adult v1.0 - Pain Interference 4a T Score | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of pain interference with daily activities. Min T Score = 41.6; Max T Score = 75.6. Raw scores are summed, then converted to T Scores from a lookup table. Higher T scores represent a worse outcome (i.e., greater pain interference).
PROMIS Pain Intensity | 1 week; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Self-report measure of average pain intensity. One item 0-10 numeric rating scale. Min score = 0, Max score = 10. Higher score represents worse outcome (i.e., greater pain intensity)
Patient Global Impression of Improvement (PGI-I) | This item assess how the patient is "right now" compared to beginning treatment; Administered at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and 3- and 6-month follow-up
  Single item self-report measure of patient perception of improvement in their urinary symptoms compared to before treatment. Rating scale from 1 (very much better) to 7 (very much worse). Lower score represents better outcome (i.e., more improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Taple BJ, Griffith JW, Weaver C, Kenton KS. Enhancing behavioral treatment for women with pelvic floor disorders: Study protocol for a pilot randomized controlled trial. Contemp Clin Trials Commun. 2020 Jan 3;17:100514. doi: 10.1016/j.conctc.2019.100514. eCollection 2020 Mar. PMID 31956723

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03623880/Prot_SAP_005.pdf
  • Informed Consent Form (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03623880/ICF_004.pdf